CLINICAL TRIAL: NCT06549959
Title: An Open-label, Randomized, Parallel Group, Single Dose Study to Investigate the Pharmacokinetics of Telitacicept Pre-filled Injection and Freeze-dried Powder Injection in Chinese Healthy Subjects
Brief Title: A Single Dose Study to Investigate the Pharmacokinetics (PK) of Telitacicept Pre-filled Injection and Freeze-dried Powder Injection in Chinese Healthy Subjects
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: RemeGen Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 18C033
Record Dates: First submitted 2024-08-06; First posted 2024-08-12 (Actual); Last update posted 2024-08-12 (Actual); Status verified 2024-08

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Telitacicept Pre-filled Injection 80mg (Experimental)
  Interventions: Drug: Telitacicept Pre-filled Injection 80mg
- Telitacicept Freeze-dried powder Injection 80mg (Experimental)
  Interventions: Drug: Telitacicept Freeze-dried powder Injection 80mg

INTERVENTIONS:
Drug: Telitacicept Pre-filled Injection 80mg — The patient received one treatment of Telitacicept 80mg in the test group
  Arms: Telitacicept Pre-filled Injection 80mg
Drug: Telitacicept Freeze-dried powder Injection 80mg — The patient received one treatment of Telitacicept 80mg in the test group
  Arms: Telitacicept Freeze-dried powder Injection 80mg

SUMMARY:
This is an open-label, randomized, parallel group, single dose study in healthy Chinese subjects. The purpose of this study is to evaluate the Pharmacokinetics and safety of Telitacicept Pre-filled Injection and Freeze-dried powder Injection.

ELIGIBILITY:
Inclusion Criteria:

1. 18-50 years old at the time of signing the informed consent form，gender is unlimited；
2. Male Weight 55-70 kg, female Weight 50-65 kg, and BMI ranging from 18 to 28 kg/m2 (including critical values);
3. Physical examination, vital signs, chest radiographs, ECG, epidemiologic tests, routine blood tests, blood biochemistry, lipids, urinalysis, and coagulation are normal，or abnormal by the investigator as having no clinical significance；
4. Fully understand the purpose and requirements of this trial, voluntarily participate in the clinical trial and sign the written informed consent, and be able to complete all trial procedures according to the trial requirements.

Exclusion Criteria:

1. Site staff and family members directly involved in the trial; or sponsor staff and family members directly involved in the implementation of the trial;
2. History of any of any nervous system, cardiovascular system, digestive system, respiratory system, urinary system, blood and lymphatic system, skeletal muscle system, immune system, metabolic system disease, or other diseases that are not suitable for clinical trials (such as mental history, malignant tumors, etc.);
3. History of lymphoproliferative disease (e.g., EB virus associated lymphoproliferative disease), lymphoma, leukemia, myeloproliferative disease, multiple myeloma, or signs and symptoms suggestive of lymphoproliferative disease;
4. History of abnormal bleeding or coagulation disorders (such as prone to bruising, gingival bleeding, prolonged bleeding after tooth extraction, joint hemorrhage, heavy menstruation leading to anemia within 1 year, postpartum hemorrhage, vitamin K deficiency, hemorrhagic disease caused by acquired coagulation factor antibodies, bleeding after trauma or surgery, etc.) , or abnormal laboratory coagulation parameters, or an inherited tendency to bleed or have coagulation dysfunction, or have a history of blood clots or bleeding, or require long-term use of anticoagulants or antiplatelet aggregation drugs;
5. During screening, 12-lead ECG showing QTcF≥450 ms in male or QTcF≥470 ms in female, or the presence of degree II/III atrioventricular block, or other clinically significant ECG abnormalities are judged by investigators not inappropriate;
6. The first-degree relatives of the subject had inherited immunodeficiency;
7. Current allergic disease, or history of allergy to therapeutic or diagnostic protein products ,allergy to alcohol(alcohol is used to sterilize injection sites), or allergy to two or more drugs and/or non-drug factors;
8. Surgery within 6 months prior to screening, or planned surgery during the trial, or within 2 weeks of the end of the trial(including cosmetic surgery, dental surgery, oral surgery, etc.);
9. Participation in a clinical trial of another drug within 3 months prior to screening;
10. Use of drugs that inhibit or induce hepatic metabolism within 4 weeks prior to randomization or need for use during the trial(e.g., inducers--barbiturates, carbamazepine, phenytoin, glucocorticoids, omeprazole; inhibitors--SSRI antidepressants, cimetidine, Diltiazem macrolides, nitroimidazoles, sedatives and hypnotics, verapamil, fluoroquinolones, antihistamines);
11. Current use of any prescription or over-the-counter (herbal, vitamins, or healthcare products). Current use is defined as use within 14 days or PK equivalent of 5 half-lives prior to randomization, whichever is longer;
12. History of Bleeding or donated more than 100ml blood 3 months before screening period, or plan to denote blood within 1 month after the trial;
13. Positive breath test results for alcohol or alcoholism in the 6 months prior to the screening period(≥14 units of alcohol per week: one standard unit contains 14g of alcohol, equals to 360ml of beer, 45ml of 40% liquor or 150ml of wine), or unable to stop drinking during the trial;
14. More than 5 cigarettes per day within 6 months prior to screening , or unable to quit smoking during the trial;
15. Consume excessive caffeine-containing beverages, foods that may affect drug metabolism within four weeks prior to screening: coffee (≥1100 mL per day), tea (≥2200 mL per day), cola (≥2200 mL per day), energy drinks (≥1100 mL per day), chocolate (≥510 g per day);
16. History of drug abuse, drug dependence, or drug use within 5 years prior to screening；
17. Subject may use weight-loss medications, or excessive dieting, or overeating during the trial;
18. Tattoos, scarring, or other conditions in the planned injection site area (front of thigh) that may interfere with the evaluation of the injection site;
19. COVID-19 vaccine within 2 weeks prior to randomization，or live vaccine within 30 days prior to randomization， or live vaccine required during the trial;
20. Positive test for Hepatitis B surface antigen (HBsAg), hepatitis C virus (HCV) antibody, human immunodeficiency virus (HIV) antibody, Treponema pallidum antibody, tuberculin test (IGRAs);
21. History of any clinically significant infections within 6 months prior to screening (e. g., requiring hospitalization or parenteral antimicrobial therapy or opportunistic infections);
22. History of symptomatic herpes zoster or herpes simplex, more than one episode of localized herpes zoster, or disseminated herpes zoster (single episode) within 12 weeks prior to screening；
23. Female subjects with a positive pregnancy test during screening period，or lactating female ; subjects and their partners do not agree to take effective contraceptive measures (such as intrauterine devices, contraceptives or condoms) throughout the trial and within 4 months after injection of the Investigational drug;
24. Investigators believe that there are other factors that are not suitable for participating in the experiment.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 248 (Estimated)
Dates: Start 2024-08-05 (Actual); Primary Completion 2024-11-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
C-max | Day 0#Day 1#Day 2#Day 3#Day 5#Day 8#Day 15#Day 22#Day 29#Day 43#Day 57
  Maximum observed plasma concentration
AUC0-∞ | Day 0#Day 1#Day 2#Day 3#Day 5#Day 8#Day 15#Day 22#Day 29#Day 43#Day 57
  Area under the plasma concentration time curve from time 0 to the time of last observed quantifiable concentration

SECONDARY OUTCOMES:
T-max | Day 0#Day 1#Day 2#Day 3#Day 5#Day 8#Day 15#Day 22#Day 29#Day 43#Day 57
  Time to reach maximum observed plasma concentration
Evaluation of AEs (adverse events) | Up to Day 57
  Through observing number of total AEs and number of subjects with AEs and other factors of AEs #to evaluate the safety and tolerance of healthy subjects.

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - The Affiliated Hospital of Guizhou Medical University, Guiyang, Guizhou
  - West China Hospital of Sichuan University, Chengdu, Sichuan
  - Tianjin People's Hospital, Tianjin, Tianjin Municipality